CLINICAL TRIAL: NCT05447533
Title: Frail Old Patients With Clostridioides Difficile Infection: Improvement of Quality in Treatment and Care
Brief Title: Clostridioides Difficile and Frailty
Acronym: CLODIFRAIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Horsens Hospital (Other); Randers Regional Hospital (Other); Central Jutland Regional Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1106
Record Dates: First submitted 2022-06-28; First posted 2022-07-07 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-05

CONDITIONS: Frail Elderly; Clostridioides Difficile; Geriatric Assessment; Faecal Microbiota Transplantation; Aged
MeSH Terms: interventions — Geriatric Assessment; Fecal Microbiota Transplantation; Standard of Care

STUDY DESIGN:
Intervention Model Description: Parallel-group randomised clinical trial (RCT). The study compares two well-known organisations of care and does not involve experimental treatments or sampling of biological material outside of routine care. It is therefore classified as a quality improvement project by the Central Denmark Region Committees on Health Research Ethics (case number 1-10-72-1-21).
Who Masked: Outcomes Assessor
Masking Description: Functional capacity and Overall Quality of life will be performed on both groups by a trained blinded project assistant during planned visits to the patients. The project assistant will be blinded to randomization status in redcap database.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Geriatric tailored assessment and intervention (Other): The geriatric tailored intervention consists of the following components:
  1. Comprehensive Geriatric Assessment
  2. Continued geriatric care during 8 weeks follow-up or until cured.
  Interventions: Other: Comprehensive geriatric assessment (CGA); Other: Continued geriatric care; Other: Faecal microbiota transplantation (FMT)
- Standard care (Active Comparator): Standard care: Patients are not contacted by the geriatric team. They receive usual treatment at the treating physician's discretion. Standard care of Clostridioides difficile infection in Denmark is described in the National clinical guideline.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Comprehensive geriatric assessment (CGA) — Within 5 weekdays from date of randomization (not included) a standardized CGA with a tailor-made intervention will be performed in the allocated ward or at home by a geriatric team. Bedside Multidimensional Prognostic Index (MPI) will be performed.
  A geriatric Clostridioides difficile infection checklist will be performed by local geriatrician and secure an early assessment of CDI and treatment strategy.
  When indication: pre-treatment with vancomycin 125 mg x 4. Routine biochemical analyses for patients with Clostridioides difficile infection.
  Evaluation of indication for faecal microbiota transplantation (FMT).
  Criteria for FMT rely on the geriatric assessment and will be considered for the patient if the patient fulfil one of the following:
  1. Severe index, recurrent or refractory CDI as defined by national clinical guidelines or
  2. High risk patient according to CGA at first visit. High risk patient is defined frailty grade MPI-2 (moderate) or MPI-3 (severe).
  Arms: Geriatric tailored assessment and intervention
Other: Continued geriatric care — Continued specialized geriatric care through 8 weeks of follow-up. Minimum of follow-up is 8 weeks from last FMT or start of vancomycin/fidaxomicin treatment.
  Tailormade telephone contacts and/or visits in case of clinical exacerbation. Performed by local geriatric teams.
  The geriatric department remains responsible for the CDI during 8 weeks of follow-up or until cured.
  Arms: Geriatric tailored assessment and intervention
Other: Faecal microbiota transplantation (FMT) — When clinical indication for FMT, this will be delivered as 15-25 capsules (~ 50 grams of donor faeces from one thoroughly screened healthy donor). If the patient is not admitted to hospital, FMT will be de-livered as home treatment via regional geriatric team or project manager and project nurse. If the patient has dysphagia diagnosed by dysphagia screening or carries a nasogastric tube, vancomycin and FMT can be delivered by naso-jejunal tube (Bengmark 10 Fr, Nutricia), requiring a referral to the Radiology department for verification of duodenal/jejunal tube placement. If available in the specific department, placement can be controlled via mobile x-ray.
  Arms: Geriatric tailored assessment and intervention
Other: Standard care — Standard care: Patients are not contacted by the geriatric team. They receive usual treatment at the treating physician's discretion.
  Arms: Standard care

SUMMARY:
CDI is a major cause of antibiotics-associated diarrhoea. More than half of the patients affected are 70 years or older and frail. Mortality among older patients with CDI is high. Faecal microbiota transplantation (FMT) is a life-saving therapy which reduce symptom duration and mortality. The FMT procedure usually requires hospital attendance, and frail old patients often are too weak to tolerate transportation to hospital and may therefore be withheld treatment.

The overall aim of the present project is to investigate whether a multimodal geriatric assessment, treatment and follow-up of frail older patients with CDI can improve patient survival compared with standard care. In particular, it is explored whether an expanded collaboration between the geriatric wards, early clinical assessment and home treatment with FMT contribute to increased patient survival rates.

DETAILED DESCRIPTION:
This is a multi-centre randomised clinical trial that test two established care pathways in the assessment and treatment of old patients with Clostridioides difficile infection (CDI). We aim to include 216 patients aged 70 years or older with Clostridioides difficile infection. Patients are randomised in a 1:1 ratio to either geriatric tailored intervention or standard care as defined by national clinical guidelines. The primary outcome is 90-day survival.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 70 years and living in the Central Denmark Region
2. Positive PCR test Clostridioides difficile

Exclusion Criteria:

1. Previously included
2. > 4 episodes of CDI
3. FMT treatment 8 weeks before date of positive PCR test for Clostridioides difficile.
4. End of life care defined as follows: end of life care treatment has been initiated before positive PCR test for CDI and the patient has days/few weeks of survival (investigator consensus based on review of electronic medical journal (EMR))
5. Patients already received Comprehensive Geriatric Assessment, defined as follows: when diagnosed with CDI affiliated with the Department of Geriatrics (in- or outpatient activity).

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 217 (Actual)
Dates: Start 2022-09-16 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-08-16 (Actual)

PRIMARY OUTCOMES:
90-day mortality | Date of 90-day follow-up will include day of positive PCR test for CD and day 90 from date of positive PCR test for CD.
  Mortality within 90 days from date of positive Polymerase Chain Reaction (PCR) test for Clostridioides difficile (CD). Date of death will be collected from the electronic medical journals according to date of death registration.

SECONDARY OUTCOMES:
Physical functional status | 83-97 weekdays after date of positive PCR test for Clostridioides difficile.
  Functional Recovery Score (FRS). Sum-score, range 100-0 (100 is the highest physical functional status score possible, 0 is the lowest).
  FRS will be performed on both groups by a blinded and trained project assessor during planned visits to the patients at 90-days follow-up. FRS will be performed according to the functional capacity at 90-day of follow-up as well as a retrospective FRS assessment according to functional capacity on the date of positive PCR test for Clostridioides difficile.
  This will be performed by asking the patient/relatives about the functional capacity. FRS will be performed within 83-97 weekdays after date of positive PCR test for Clostridioides difficile.
Overall quality of life assessed by Depression List | 83-97 weekdays after date of positive PCR test for Clostridioides difficile.
  The Overall quality of life will be assessed by the Overall Quality of Life Depression List (OQoL-DL) and will be performed on both groups by a blinded and trained project assessor during planned visits to the patients at 90-days follow-up within 83-97 weekdays after date of positive PCR test for Clostridioides difficile.
Quality of life assessed by the 5-level EQ-5D Interviewer version | 83-97 weekdays after date of positive PCR test for Clostridioides difficile.
  The quality of life will be assessed by the 5-level EQ-5D version (EQ-5D-5L). The EQ-5D-5L be performed on both groups by a blinded and trained project assessor during planned visits to the patients at 90-days follow-up within 83-97 weekdays after date of positive PCR test for Clostridioides difficile.
Quality of life assessed by the 5-level EQ-5D proxy 2 version | 83-97 weekdays after date of positive PCR test for Clostridioides difficile.
  The quality of life will be assessed by the 5-level EQ-5D proxy 2 version (EQ-5D-5L). The EQ-5D-5L proxy 2 version be performed in both groups by proxy invited online. The significant others (proxy) will receive the survey at 90-days follow-up within 83-97 weekdays after date of positive PCR test for Clostridioides difficile.

OTHER OUTCOMES:
Recurrent Clostridioides difficile infection | Within period of 90-day follow-up from date of positive PCR test for Clostridioides difficile.
  Recurrent CDI is defined as a new CDI episode after ended treatment for CDI with treatment response. New episode of diarrhea (≥3 loose stools, Bristol 6-7) and a positive Clostridioides difficile PCR test. Outcome will be collected from electronic medical journals.
Time to Faecal microbiota transplantation | Within period of 90-day follow-up.
  Time from date of positive PCR test for Clostridioides difficile to date of faecal microbiota transplantation.
Time to initiation of vancomycin/bactocin treatment | Within period of 90-day follow-up.
  Time from positive PCR test for Clostridioides difficile to date of initiation of medical treatment with vancomycin/bactocin.
Readmission in patients diagnosed with Clostridioides difficile during hospitalisation | Within a period of 30 days after hospital discharge.
  Readmission defined as any unplanned, acute rehospitalisation (elective or planned admissions and outpatient procedures excluded) at any hospital within the Central Denmark Region, occurring within four hours from index admission and up to 30 days after hospital discharge.
Days in hospital | Within period of 90-day follow-up after positive PCR test for CD.
  Number of days in hospital from date of positive PCR test for CD and until 90 days.

CONTACTS AND LOCATIONS:
Overall Officials: Else Marie Damsgaard, Professor, Principal Investigator — Department of Geriatrics, Aarhus University Hospital
Locations (1):
- Department of Geriatrics, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bauer MP, Notermans DW, van Benthem BH, Brazier JS, Wilcox MH, Rupnik M, Monnet DL, van Dissel JT, Kuijper EJ; ECDIS Study Group. Clostridium difficile infection in Europe: a hospital-based survey. Lancet. 2011 Jan 1;377(9759):63-73. doi: 10.1016/S0140-6736(10)61266-4. PMID 21084111
- [Background] Czepiel J, Krutova M, Mizrahi A, Khanafer N, Enoch DA, Patyi M, Deptula A, Agodi A, Nuvials X, Pituch H, Wojcik-Bugajska M, Filipczak-Bryniarska I, Brzozowski B, Krzanowski M, Konturek K, Fedewicz M, Michalak M, Monpierre L, Vanhems P, Gouliouris T, Jurczyszyn A, Goldman-Mazur S, Wultanska D, Kuijper EJ, Skupien J, Biesiada G, Garlicki A. Mortality Following Clostridioides difficile Infection in Europe: A Retrospective Multicenter Case-Control Study. Antibiotics (Basel). 2021 Mar 13;10(3):299. doi: 10.3390/antibiotics10030299. PMID 33805755
- [Background] Cober ED, Malani PN. Clostridium difficile infection in the "oldest" old: clinical outcomes in patients aged 80 and older. J Am Geriatr Soc. 2009 Apr;57(4):659-62. doi: 10.1111/j.1532-5415.2009.02182.x. PMID 19392957
- [Background] Hensgens MP, Goorhuis A, Dekkers OM, van Benthem BH, Kuijper EJ. All-cause and disease-specific mortality in hospitalized patients with Clostridium difficile infection: a multicenter cohort study. Clin Infect Dis. 2013 Apr;56(8):1108-16. doi: 10.1093/cid/cis1209. Epub 2013 Jan 8. PMID 23300235
- [Background] Ellis G, Gardner M, Tsiachristas A, Langhorne P, Burke O, Harwood RH, Conroy SP, Kircher T, Somme D, Saltvedt I, Wald H, O'Neill D, Robinson D, Shepperd S. Comprehensive geriatric assessment for older adults admitted to hospital. Cochrane Database Syst Rev. 2017 Sep 12;9(9):CD006211. doi: 10.1002/14651858.CD006211.pub3. PMID 28898390
- [Background] Gregersen M, Pedersen AB, Damsgaard EM. Comprehensive geriatric assessment increases 30-day survival in the aged acute medical inpatients. Dan Med J. 2012 Jun;59(6):A4442. PMID 22677240
- [Background] Leibovici-Weissman Y, Atamna A, Schlesinger A, Eliakim-Raz N, Bishara J, Yahav D. Risk factors for short- and long-term mortality in very old patients with Clostridium difficile infection: A retrospective study. Geriatr Gerontol Int. 2017 Oct;17(10):1378-1383. doi: 10.1111/ggi.12866. Epub 2016 Sep 20. PMID 27647625
- [Background] Jorgensen SMD, Rubak TMM, Damsgaard EM, Dahlerup JF, Hvas CL. Faecal microbiota transplantation as a home therapy to frail older people. Age Ageing. 2020 Oct 23;49(6):1093-1096. doi: 10.1093/ageing/afaa073. PMID 32365381
- [Background] Hvas CL, Dahl Jorgensen SM, Jorgensen SP, Storgaard M, Lemming L, Hansen MM, Erikstrup C, Dahlerup JF. Fecal Microbiota Transplantation Is Superior to Fidaxomicin for Treatment of Recurrent Clostridium difficile Infection. Gastroenterology. 2019 Apr;156(5):1324-1332.e3. doi: 10.1053/j.gastro.2018.12.019. Epub 2019 Jan 2. PMID 30610862
- [Derived] Rubak T, Baunwall SMD, Gregersen M, Paaske SE, Asferg M, Barat I, Secher-Johnsen J, Riis MG, Rosenbaek JB, Hansen TK, Orum M, Steves CJ, Veilbaek H, Hvas CL, Damsgaard EMS. Early geriatric assessment and management in older patients with Clostridioides difficile infection in Denmark (CLODIfrail): a randomised trial. Lancet Healthy Longev. 2024 Dec;5(12):100648. doi: 10.1016/j.lanhl.2024.100648. Epub 2024 Oct 30. PMID 39488230

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-06-26): https://cdn.clinicaltrials.gov/large-docs/33/NCT05447533/SAP_000.pdf